CLINICAL TRIAL: NCT07357467
Title: Effect of Oral Supplement Intervention on Influenza Vaccine Long-term Efficacy: a Follow-up Study
Brief Title: Effect of Oral Supplement on Influenza Vaccine Long-term Response
Acronym: EOSIIVE-F
Status: Not yet recruiting | Type: Observational
Sponsor: Tsinghua University (Other)
Collaborators: Second Affiliated Hospital of Bengbu Medical College (Other)
Responsible Party: Principal Investigator, Ai Zhao, Associate Professor, Tsinghua University
Other Study IDs: THU01-20251109
Record Dates: First submitted 2026-01-12; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Influenza; Immunosenescence
Keywords: Tauroursodeoxycholic Acid (TUDCA); Influenza Vaccine; Antibody; Memory B Cells; Long-lived Plasma Cells; Elderly Adults; Humoral Immunity; Nutritional Immunomodulation; Bile Acids
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TUDCA Supplementation Group: Participants who received TUDCA supplementation (1000 mg/day) during the original study (February-April 2025). In the original trial, participants took 1000 mg of TUDCA (Tauroursodeoxycholic acid) dietary supplement capsules daily. Each capsule contained 500 mg of TUDCA (two capsules per serving). Participants maintained their usual lifestyle during the intervention: Day 0-Day 2 served as an adaptation period; on Day 3, they received a quadrivalent influenza vaccine, followed by continued supplementation until Day 24. This extended follow-up study involves no intervention, only a single fasting blood draw (20 mL) approximately 12 months post-vaccination to assess long-term immune responses.
- Placebo Group: Participants who received placebo during the original study (February-April 2025). In the original trial, participants took placebo capsules identical in appearance and smell to the TUDCA capsules. Participants maintained their usual lifestyle during the intervention: Day 0-Day 2 served as an adaptation period; on Day 3, they received a quadrivalent influenza vaccine, followed by continued placebo supplementation until Day 24. This extended follow-up study involves no intervention, only a single fasting venous blood draw (approximately 20 mL) about 12 months post-vaccination to assess long-term immune responses.

SUMMARY:
This is a follow-up study of a previously completed randomized controlled trial (NCT06827873) that investigated the effects of oral supplements on influenza vaccine response in adults aged 60-70 years. The original study was completed in April 2025, with participants receiving either TUDCA (Tauro Ursodesoxy Cholic Acid) supplementation, fatty acid supplementation, or placebo during influenza vaccination.

The primary objectives of this follow-up study are to:

1. Evaluate the durability of vaccine-induced antibody responses approximately 8 months post-vaccination
2. Assess the persistence of immune memory cells, particularly long-lived plasma cells and memory B cells
3. Compare long-term immune responses between the TUDCA supplementation group and placebo group

This observational follow-up involves a single visit where participants will:

1. Provide one blood sample for antibody and immune cell analysis
2. No intervention or vaccination will be administered

The study will specifically focus on B cell subsets through flow cytometry analysis, including total B cells, memory B cells, plasma cells, and long-lived plasma cells. This research aims to determine whether TUDCA supplementation can enhance the durability of vaccine-induced immunity in older adults.

DETAILED DESCRIPTION:
Influenza virus infection presents a significant global health challenge, particularly threatening the elderly population due to immunosenescence. The immune response to influenza vaccination involves a complex series of events: after vaccination, hemagglutination inhibition antibody titers peak around day 14, accompanied by the production of neutralizing antibodies and other specific antibodies. This immune response gradually stabilizes to a post-response baseline level as immune memory establishes.

The age-related decline in immune function manifests through multiple mechanisms, including: reduced production of naive T cells; decreased diversity of T cell repertoire; compromised B cell function; and altered cytokine production profiles, which all diminish vaccine response efficacy. Recent advances in immunometabolism have revealed the crucial role of specific fatty acids and bile acids in immune system modulation. Our preliminary explorations found that fatty acid intervention could significantly reduce the time required for antibody production and enhance its levels following rabies vaccination. We also noticed that serum Tauroursodeoxycholic Acid (TUDCA) was elevated in the intervention group. However, the related mechanisms remain unclear.

Besides, evidence from influenza vaccine studies reveals critical temporal dynamics: antibody titers peak at 1-1.3 months post-vaccination, decline by 3 months, yet remain elevated above baseline at 6 months. Vaccine effectiveness demonstrates time-dependent reduction from 80% at 14 days to 37% at 128 days and 46% at 180 days post-vaccination. Crucially, antibody persistence correlates with long-lived plasma cells (LLPCs), which maintain continuous antibody secretion, while memory B cells enable rapid secondary responses upon antigen re-exposure by differentiating into plasma cells and LLPCs.

Building on these findings, we hypothesized that TUDCA itself may play an active immunoregulatory role during vaccination, influencing B-cell differentiation and antibody persistence. To test this hypothesis and further characterize its potential benefits in elderly populations, we designed an extended follow-up study.

The original study (February-April 2025) demonstrated that TUDCA supplementation significantly enhanced memory B cell responses compared to placebo and fatty acid supplementation groups during the acute phase post-vaccination (Day 0-24). In this extended follow-up, conducted approximately 12 months after vaccination, participants will return for a single fasting venous blood draw (approximately 10 mL) to assess antibody titers and characterize immune-cell subsets. No further intervention or vaccination will be performed. This timepoint represents a critical window for assessing immune durability in the elderly. By quantifying long-term antibody titers and characterizing B cell subsets-particularly plasma cells and long-lived plasma cells-we will determine whether TUDCA supplementation enhances the persistence of vaccine-induced humoral and cellular immunity. This investigation addresses whether nutritional strategies can extend vaccine protection duration in older adults, where immunosenescence substantially limits both vaccine efficacy and protection longevity.

ELIGIBILITY:
Inclusion Criteria:

1. Originally assigned to either the TUDCA supplementation group or placebo control group
2. No influenza vaccination or other vaccines received between April 2025 and December 2025
3. Willing to participate in this follow-up study and sign supplementary informed consent
4. Stable health condition

Exclusion Criteria:

1. Started using immunosuppressants or hormonal medications after the original study
2. Experienced serious illness or hospitalization within the past month, or planning surgery soon
3. Experienced fever, cold, severe diarrhea, or taken influenza antiviral medications within the past month
4. Unable or unwilling to participate in blood collection
5. Lost to follow-up or unable to contact

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This extended follow-up study includes participants from the original randomized controlled trial (Protocol ID: THU01-20240201; NCT06827873) conducted between February and April 2025. Thirty older adults (aged 60-70 years) were previously randomized to either the TUDCA group (n=15) or placebo group (n=15). All completed the 25-day intervention, received quadrivalent influenza vaccine on Day 3, and finished all Day 24 assessments. Participants were recruited from community health centers affiliated with the Second Affiliated Hospital of Bengbu Medical College, Anhui, China, and provided written informed consent for both the original and follow-up studies.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Long-term Influenza-Specific Antibody Levels Post-Vaccination | Day 360 (approximately 12 months post-vaccination)
  Evaluate influenza virus-specific IgG antibody levels at approximately 12 months post-vaccination to assess the durability of vaccine-induced humoral immunity. Antibody levels will be measured for all four strains contained in the quadrivalent influenza vaccine (H1N1, H3N2, B/Victoria, B/Yamagata) using ELISA or hemagglutination inhibition (HI) assay.

SECONDARY OUTCOMES:
B Cell Immune Memory Persistence | Day 360 (approximately 12 months post-vaccination)
  Assess B cell subsets through flow cytometry analysis, including Total B cells (CD19+), Memory B cells (CD19+ & CD27+), Plasma cells (CD19+, CD38+ & CD27+) and Long-lived plasma cells (CD19+, CD38+ & CD138+). Compare the persistence of these immune memory cell populations between TUDCA supplementation and placebo groups to evaluate whether TUDCA enhances long-term cellular immunity.

OTHER OUTCOMES:
Safety Assessment | Day 360 (at blood collection visit, 12 months post-vaccination)
  Record and monitor any adverse events related to blood collection, including pain, dizziness, bruising, or hematoma formation. In addition, participants will be asked to report any delayed or persistent adverse effects that may have occurred since completion of the original study, including those potentially associated with prior vaccination or nutritional supplementation. These events will be documented and evaluated descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Cong Tian, Master, Study Director — The Second Affiliated Hospital of Bengbu Medical College
Locations (1):
- Tsinghua University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mordant FL, Price OH, Rudraraju R, Slavin MA, Marshall C, Worth LJ, Peck H, Barr IG, Sullivan SG, Subbarao K. Antibody titres elicited by the 2018 seasonal inactivated influenza vaccine decline by 3 months post-vaccination but persist for at least 6 months. Influenza Other Respir Viruses. 2023 Jan;17(1):e13072. doi: 10.1111/irv.13072. Epub 2022 Nov 30. PMID 36451293
- [Background] Ellebedy AH. Immunizing the Immune: Can We Overcome Influenza's Most Formidable Challenge? Vaccines (Basel). 2018 Sep 22;6(4):68. doi: 10.3390/vaccines6040068. PMID 30248996
- [Background] Ferdinands JM, Fry AM, Reynolds S, Petrie J, Flannery B, Jackson ML, Belongia EA. Intraseason waning of influenza vaccine protection: Evidence from the US Influenza Vaccine Effectiveness Network, 2011-12 through 2014-15. Clin Infect Dis. 2017 Mar 1;64(5):544-550. doi: 10.1093/cid/ciw816. Epub 2016 Dec 29. PMID 28039340